CLINICAL TRIAL: NCT02020876
Title: GenomeDx Decipher Test for Metastatic Disease in Prostate Cancer for Patients With Adverse Pathology Post Radical Prostatectomy: Does it Impact Physician Decision Making?
Brief Title: Decision Impact Study to Measure the Influence of DECIPHER on Treatment Recommendations
Acronym: DECIDE
Status: Completed | Type: Observational
Sponsor: GenomeDx Biosciences Corp (Industry)
Responsible Party: Sponsor
Other Study IDs: CU001
Record Dates: First submitted 2013-12-18; First posted 2013-12-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Practicing urologic surgeons: Performing at least 60 radical prostate surgeries annually
  Interventions: Other: DECIPHER Questionnaire

INTERVENTIONS:
Other: DECIPHER Questionnaire — Participants are asked to complete a questionnaire to assess the impact of Decipher on physicians' treatment recommendation. All participants use the same data collection instrument. Each participant opinion is collected based on a random selection of cases.

SUMMARY:
This clinical utility study pilot is based on a review of real but de-identified and randomized patient cases and aims to evaluate Urologists' treatment recommendations before and after reviewing the results provided by the Decipher test. This is a pilot study and the primary intent is to help guide development and design of future clinical utility studies for Decipher

DETAILED DESCRIPTION:
The primary and secondary objectives will be assessed in retrospectively selected prostate cancer patients treated with radical prostatectomy with one or more adverse pathological features (APFs)

ELIGIBILITY:
Criteria (Participant enrollment)

Inclusion Criteria Study participants:

1. Practicing board-certified urologic surgeons
2. Performing at least 40 radical prostate surgeries annually

Exclusion Criteria Study Participants:

(1) Did not meet the inclusion criteria

Criteria (Case selection)

Inclusion Criteria Case File:

Patient cases eligible for this study were treated with radical prostatectomy and have one or more adverse pathological features present defined as:

Pathological Gleason score >= 8 or Gleason score 7 with primary pattern 4; Pathological stage T3A (= Extraprostatic extension) or T3B (=Seminal vesicle invasion); Positive surgical margins Gleason grade upgrade from biopsy to surgery

Exclusion Criteria Case File:

Metastatic disease (M+) prior to surgery Received any neo-adjuvant prostate cancer treatment with radical prostatectomy (radiation, hormone, chemotherapy)

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is an exploratory study utilizing archived tumor specimens and demographic and pathologic characteristics derived from the patient's medical charts. The study participants are the urologists who review the selected case files.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in treatment recommendation | 1.5 years
  To determine the extent to which the use of the Decipher test influences treatment recommendations by physicians post radical prostatectomy (RP).
  This decision impact study aims to evaluate Urologists' treatment recommendations before and after reviewing the results provided by the Decipher test.

SECONDARY OUTCOMES:
Urologist's perception regarding the utility of the Decipher | 1.5 years
  * Changes in Urologists expressed level of confidence in the treatment recommendation as measured by the response to item 4a in the eCRF survey.
  * Urologist's perception regarding the utility of the Decipher test as measured by the responses to question 4b and 38b and 38c in the eCRF survey.
  * Agreement in treatment recommendation

CONTACTS AND LOCATIONS:
Overall Officials: Elai Davicioni, pHd, Principal Investigator — GenomeDx Biosciences Inc.; Badani Ketan, MD, Principal Investigator — Department of Urology, Columbia University, New York, NY USA
Locations (1):
- GenomeDx Bioscience Inc., San Diego, California, United States

REFERENCES:
- [Result] Badani K, Thompson DJ, Buerki C, Davicioni E, Garrison J, Ghadessi M, Mitra AP, Wood PJ, Hornberger J. Impact of a genomic classifier of metastatic risk on postoperative treatment recommendations for prostate cancer patients: a report from the DECIDE study group. Oncotarget. 2013 Apr;4(4):600-9. doi: 10.18632/oncotarget.918. PMID 23592338